CLINICAL TRIAL: NCT04848623
Title: Identification of Vocal Biomarkers to Monitor the Health of People with a Chronic Disease
Acronym: CoLive Voice
Status: Recruiting | Type: Observational
Sponsor: Luxembourg Institute of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: CoLive Voice
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Chronic Disease
Keywords: vocal biomarker; digital biomarker; digital health; artificial intelligence; telemonitoring; medical devices; precision health digital biomarker
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The CoLive Voice research project aims to identify vocal biomarkers of severe conditions and frequent health symptoms. The project is based on digital technologies and statistical algorithms. This is an international anonymous survey where vocal recordings are collected simultaneously with large validated clinical and epidemiological data, in the context of various chronic diseases or frequent health symptoms in the general population.

DETAILED DESCRIPTION:
With the objective of using vocal biomarkers for diagnosis, risk prediction/stratification and remote monitoring of various clinical outcomes and symptoms, there is a major need to develop surveys where audio data and clinical, epidemiological and patient-reported outcomes data are collected simultaneously.

The objectives of CoLive Voice are:

* To launch an international anonymized survey where vocal recordings are associated with large validated clinical and epidemiological data, in the context of various chronic diseases or frequent health symptoms in the general population
* To extract audio features and train supervised machine learning models to identify key candidate vocal biomarkers of the aforementioned chronic conditions or related symptoms.

Participants will be recruited online and will complete the survey using a web application.

They will first answer a detailed questionnaire on their health status and then do 5 different voice records:

1. read a 30 sec prespecified text (from the Human Rights Declaration),
2. sustain voicing the vowel /aaaaaa/ as long and as steady as they can at a comfortable loudness
3. cough 3 times
4. breath in and out deeply 3 times
5. Count from 1 to 20 at a normal speed

Vocal records will be pre-processed and converted into features, meaning the most dominating and discriminating characteristics of a vocal signal. Following the selection of features, machine or deep learning algorithms will be trained to automatically predict or classify the clinical, medical or epidemiological outcomes of interest, from vocal features alone or in combination with other health-related data.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and adults > 15 years
* With or without health conditions
* From all countries

Exclusion Criteria:

* Children < 15 years

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult and adolescent above 15 years, regardless of their health status and their residence country.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2021-06-26 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Stress | At baseline
  Patient reported outcome

SECONDARY OUTCOMES:
Fatigue | At baseline
  Patient reported outcome using the fatigue severity scale (FSS). Minimum value =1, max value = 7 ; 7 is the highest level of fatigue
Hypertension | At baseline
  Patient reported outcome
Diabetes | At baseline
  Patient reported outcome
Migraine | At baseline
  Patient reported outcome
Covid-19 | At baseline
  Patient reported outcome
Overall pain | At baseline
  Patient reported outcome
Respiratory problems | At baseline
  Patient reported outcome
Level of quality of life | At baseline
  Patient reported outcome

CONTACTS AND LOCATIONS:
Overall Officials: Guy Fagherazzi, PhD, Principal Investigator — LIH
Locations (1):
- Luxembourg Institute of Health, Luxembourg, Luxembourg

REFERENCES:
- [Derived] Elbeji A, Pizzimenti M, Aguayo G, Fischer A, Ayadi H, Mauvais-Jarvis F, Riveline JP, Despotovic V, Fagherazzi G. A voice-based algorithm can predict type 2 diabetes status in USA adults: Findings from the Colive Voice study. PLOS Digit Health. 2024 Dec 19;3(12):e0000679. doi: 10.1371/journal.pdig.0000679. eCollection 2024 Dec. PMID 39700066